CLINICAL TRIAL: NCT01790529
Title: Randomized Controlled Trial to Evaluate the Optimal Timing of Surgical Antimicrobial Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Cantonal Hospital of Aarau, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SSI-19/12
Record Dates: First submitted 2013-02-05; First posted 2013-02-13 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Prophylaxis (Experimental): Early administration of SAP (Cefuroxime (plus metronidazole in colorectal surgery)) in anesthetic room (75 to 30 minutes prior to skin incision)
  Interventions: Procedure: Early administration of SAP (Cefuroxime (plus metronidazole in colorectal surgery)) in anesthetic room (75 to 30 minutes prior to skin incision)
- Late Prophylaxis (Active Comparator): Late administration of SAP (Cefuroxime (plus metronidazole in colorectal surgery)) in the operating theatre (within 30 minutes prior to skin incision)
  Interventions: Procedure: Late administration of SAP (Cefuroxime (plus metronidazole in colorectal surgery)) in the operating theatre (within 30 minutes prior to skin incision)

INTERVENTIONS:
Procedure: Early administration of SAP (Cefuroxime (plus metronidazole in colorectal surgery)) in anesthetic room (75 to 30 minutes prior to skin incision)
  Arms: Early Prophylaxis
Procedure: Late administration of SAP (Cefuroxime (plus metronidazole in colorectal surgery)) in the operating theatre (within 30 minutes prior to skin incision)
  Arms: Late Prophylaxis

SUMMARY:
Surgical site infections (SSI) are the most frequent hospital acquired infections in patients who underwent surgery. With regards to the increasing financial restraint in patient care, the socio-economic burden of SSI in the public health sector and its prevention gains in importance.

The prophylactic application of antibiotics (surgical antimicrobial prophylaxis, SAP) prior to the skin incision significantly reduces the risk of SSI, but the correct time point of drug administration remains unclear. Most studies recommend application of SAP directly prior to skin incision. Other studies, however, suggest that this is too late and more time between administration of the SAP and skin incision is necessary for optimal SSI prevention. A large cohort study in Switzerland concluded that SAP should be applied between 74 and 30 minutes prior to skin incision.

Due to the obvious importance of this controversy, we want to answer this question with a clinical study (randomized controlled trial, RCT) at the University Hospital of Basel and the Cantonal Hospital of Aarau. We plan to investigate two administration strategies according to the timing of the SAP. Strategy A will consist of SAP application in the anesthetic room located in front of the actual operating theatre, where the patient gets anesthesia. Therefore, the application of SAP will take place early, approximately between 75 and 30 minutes prior to skin incision. In strategy B we will apply SAP in the operating theatre, which on average occurs later (approximately within the last 30 minutes before skin incision).

We test the hypothesis that strategy A is more effective in preventing SSI than strategy B. We will include a total of 5000 patients in abdominal, vascular and trauma surgery (2500 at each study site and 2500 per study group). All patients will be followed in the hospital for SSI occurrence. Additionally, all patients will be interviewed by telephone after hospital discharge at a defined follow-up period of 30 days (1 year if an implant is in place, such as hip endoprosthesis or meshes). We expect this study to be completed within approximately 3 years.

DETAILED DESCRIPTION:
Additionally, the association between the following pre-defined variables and the occurence of SSI, mortality, morbidity and length of hospital stay (LOS) will be investigated:

* laparoscopy
* tutorial assistance during operation
* obesity (Body Mass Index, BMI)
* preoperative Virtual Reality (VR) training
* Adherence to Enhanced Recovery After Surgery (ERAS) concept
* smoking status
* perioperative blood glucose levels
* preoperative levels of HbA1c
* intensified insulin resistance as measured by Homeostasis Model Assessment (HOMA) and quantitative insulin-sensitivity check index (QUICKI)
* type of diabetes (IDDM vs. NIDDM)
* intraoperative Hypothermia (body core temperature)
* Lack of adherence to the principles of asepsis during surgery
* surgical experience
* patients age
* Malnutrition, measured by Hypalbuminaemia
* emergency operations
* immunosuppression and steroids
* Predictive value of Procalcitonin
* American Society of Anesthesiologists (ASA) classification
* intraoperative blood transfusion
* preoperative wound class

Amendments:

The following changes were made to the study protocol according to amendments approved by the local ethics committee:

* As of April 22nd, 2013, or the 222. patient randomized at the University Hospital Basel, the time the SAP infusion STARTED was recorded instead of the time that it ENDED. The decision to change this important parameter was taken in order to make results of this trial more comparable to those of other published studies.
* In the original study protocol it was planned to provide each randomized patient with a patient's diary to record signs of SSI. This was abandoned for limited benefit and in order to minimize patients' time and effort.
* Patients who undergo combined surgery (by one of the participating surgical specialties plus by a non participating specialty) shall not be included in this trial as outcomes (SSI) could be difficult to correlate to one or another part of surgery. This had not been specified as an exclusion criterion in the original study protocol.
* Patients' information sheets and informed consents in one of the languages other than German were only approved by the local ethics committees by May 15th, 2013.
* As per ethics committees regulations, patients can only be included in more than one clinical trials under specific circumstances. Therefore only a limited percentage of patients that are already included in other studies can still be included for this trial. However, overall, this only excludes a very limited number of potentially includable patients.

The following additional amendments were authorized by the ethics committees on August 9th, 2014:

- Version 4 of the patients' information and the written consent form. In these new versions, patients are specifically asked for permission to review their general practitioners' notes concerning potential SSI, for planned follow up as well as in case of readmission to hospital. This is specified in the study protocol, but had not been specifically mentioned in the patients' information and consent forms. This change is also intended to significantly decrease the number of patients lost to follow up as it proved difficult to contact some patients by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Inpatient visceral, vascular and trauma procedures
* SAP indicated according to clinical standards (CDC guidelines for surgical wound classification)
* informed consent

Exclusion Criteria:

* Contraindication for study drugs
* Pre-existing antibiotic therapy within 14 days of surgery
* Any doubt that patients can make the decision to participate fully informed due to cognitive impairment, such as in critically ill or demented patients.
* Emergency procedures with planned incision within 2 hours after the surgeon indicated the procedure
* Participation in other studies that could potentially interfere with the present one (according to the ethics committee)
* Combined surgery including surgical subspecialties other than the above mentioned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | 30 days
  Surgical Site Infection within 30 days after index surgery

SECONDARY OUTCOMES:
All-cause 30 day mortality | 30 days
Length of hospital stay | 1 year
Economic burden of SSI | 1 year
Nosocomial infections | 1 year
In-hospital complications | 1 year
  according to the Clavien-Dindo-Classification
Surgical Site Infection (SSI) | 1 year
  Surgical Site Infection within 1 year after surgery only for implant surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Walter P. Weber, MD, Principal Investigator — University Hospital Basel, Basel 4031 Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835
- [Derived] Kopp Lugli A, Marti WR, Salm L, Mujagic E, Bundi M, von Strauss M, Bucheli Laffer E, Landin J, Fux CA, Coslovsky M, Weber WP, Kindler C. The Role of HbA1c as a Positive Perioperative Predictor of Surgical Site and Other Postoperative Infections: An Explorative Analysis in Patients Undergoing Minor to Major Surgery. World J Surg. 2022 Feb;46(2):391-399. doi: 10.1007/s00268-021-06368-x. Epub 2021 Nov 8. PMID 34750659
- [Derived] Weber WP, Mujagic E, Zwahlen M, Bundi M, Hoffmann H, Soysal SD, Kraljevic M, Delko T, von Strauss M, Iselin L, Da Silva RXS, Zeindler J, Rosenthal R, Misteli H, Kindler C, Muller P, Saccilotto R, Lugli AK, Kaufmann M, Gurke L, von Holzen U, Oertli D, Bucheli-Laffer E, Landin J, Widmer AF, Fux CA, Marti WR. Timing of surgical antimicrobial prophylaxis: a phase 3 randomised controlled trial. Lancet Infect Dis. 2017 Jun;17(6):605-614. doi: 10.1016/S1473-3099(17)30176-7. Epub 2017 Apr 3. PMID 28385346
- [Derived] Mujagic E, Zwimpfer T, Marti WR, Zwahlen M, Hoffmann H, Kindler C, Fux C, Misteli H, Iselin L, Lugli AK, Nebiker CA, von Holzen U, Vinzens F, von Strauss M, Reck S, Kraljevic M, Widmer AF, Oertli D, Rosenthal R, Weber WP. Evaluating the optimal timing of surgical antimicrobial prophylaxis: study protocol for a randomized controlled trial. Trials. 2014 May 24;15:188. doi: 10.1186/1745-6215-15-188. PMID 24885132